CLINICAL TRIAL: NCT01027520
Title: Day One Post Operative Range of Motion Following Skin Graft to Hand With Intraoperative Coban Dressing
Brief Title: Range of Motion Following Intraoperative Coban Dressing Application in Hand Burns
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment numbers
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Cathy Barrow, Occupational Therapist, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cobandressing
Record Dates: First submitted 2009-12-04; First posted 2009-12-08 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2016-09

CONDITIONS: Burns; Hand Injuries
Keywords: Hand burn; skin graft; coban dressing; range of motion
MeSH Terms: conditions — Burns; Hand Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Application of Coban dressing
  Interventions: Other: application of coban dressing

INTERVENTIONS:
Other: application of coban dressing — application of a intraoperative coban dressing with reapplications following dressing removal.
  Other Names: 3M Coban Self-Adherent wrap

SUMMARY:
Participants of this study will include burns requiring skin graft to hand(s). After informed consent, an occupational therapy evaluation will be performed. Participants will consent to surgery, in which skin graft will be applied by physician during surgery, occupational therapy will apply coban dressing. Participant will seen daily by occupational therapist during hospitalization for active range of motion to hand(s). Occupational therapist will measure range of motion of hand(s) and physician will assess graft success at one and four days after surgery and at three out patient clinic visits. Hand strength will also be measured at three out patient visits.

Does the initiation of range of motion on post operative day kone with coban dressing improve hand function without compromising graft success?

DETAILED DESCRIPTION:
The participant will be evaluated by occupational therapist prior to surgery. The coban dressing will be applied to the participant's hand(s)during surgery for a skin graft. This portion will occur whether the participant agrees to participate or not. The participant will begin range of motion exercises the day after surgery (post operative day one) with and occupational therapist. The occupational therapist will see the participant daily for supervised range of motion while in the hospital. The coban dressing will be removed on post operative day one if a sheet graft is placed to assess bleeding under graft. The coban dressing will be reapplied and removed again on post operative day four. When a meshed graft is placed, coban dressing will be removed on post operative day four only. All skin grafts (meshed and sheet grafts) and range of motion will be assessed on post operative day four. Coban dressing will be reapplied. The participant will continue range of motion exercise program at home. An appointment will be scheduled for 3 consecutive weeks in out patient burn clinic. During clinic visits, skin graft, range of motion, and grip strength will be measured. The participant will seen in out patient burn clinic whether they choose to participate in the study or not as a standard of burn care.

ELIGIBILITY:
Inclusion Criteria:

* Less than 15% burn, burn requires skin graft to dorsum of hand, burn involves at least 2 metacarpophalangeal joints
* 18 and older

Exclusion Criteria:

* Latex allergy
* Documented diagnoses of mental illness that interferes with patients ability to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
hand function(range of motion, grip and pinch strength) | post operative day four, first, second and third clinic visits

SECONDARY OUTCOMES:
graft success | post operative day 4 and first, second and third clinic visits

CONTACTS AND LOCATIONS:
Overall Officials: Catherine L Barrow, BS OT, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Health Care - George David Peak Memorial Burn Center, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No